CLINICAL TRIAL: NCT05734443
Title: Effects of Task-Specific Step Training on Reactive Balance After Laboratory-Induced Trips: A Pilot Trial
Brief Title: Effects of Task-Specific Step Training on Reactive Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-1072
Record Dates: First submitted 2023-02-08; First posted 2023-02-21 (Actual); Results first posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2023-09

CONDITIONS: Accidental Fall

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- step training (Experimental): Two training sessions per week will be completed for three consecutive weeks. Each training session will last 0.5-1 hour with an active training time of 30 minutes per participant. Training will involve repeated volitional and reactive stepping movements that mimic the movements necessary to recover balance after tripping while walking.
  Interventions: Behavioral: step training
- treadmill training (Experimental): Two training sessions per week will be completed for three consecutive weeks. Each training session will last 0.5-1 hour with an active training time of 30 minutes per participant. Training will involve repeated exposure to simulated trips on a treadmill. To simulate a trip, participants first stand on the stationary treadmill belt. A sudden and unexpected increase in backward treadmill belt speed induces a forward loss of balance similar to when tripping. Participants are then required to take steps to recover balance and establish a stable gait pattern before the trial ends. Trials are repeated using pseudo-random speeds that provide variability and are individualized to each participant's capabilities.
  Interventions: Behavioral: treadmill training
- Control (No Intervention)

INTERVENTIONS:
Behavioral: step training — Participants practice volitional and reactive stepping responses that mimic those needed when recovering balance after tripping.
  Arms: step training
Behavioral: treadmill training — Sudden treadmill changes in speed (from standing) induce trip-like losses of balance, after which participants take steps to recover balance and establish a stable gait pattern. This is repeated over a range of speeds to both provide training variability and to individualize training to each participant's capability.
  Arms: treadmill training

SUMMARY:
The goal of this clinical trial is to evaluate a novel and pragmatic (i.e., not requiring specialized equipment) task-specific step training regimen that aims to improve reactive balance after tripping. The main questions it aims to answer are:

* Does this step training regimen improve reactive balance after tripping compared to no training?
* How well does this step training regimen improve reactive balance compared to treadmill training, which is a more commonly studied reactive balance training regimen that uses a specialized treadmill.

Participants will:

* complete step training or treadmill training (or no training if assigned to the control group) twice a week for three weeks
* experience a laboratory-induced trip three weeks later to evaluate their reactive balance

ELIGIBILITY:
Inclusion Criteria:

* 65-80 years old
* willing to use wearable sensors for 2-3 weeks (for a separate study)
* no lower limb amputation
* not weigh over 250 pounds
* pass a telephone interview related to cognitive status

Exclusion Criteria:

* participants must pass a health screening involving a questionnaire that will be reviewed by a health care specialist.
* participants must not have clinical osteoporosis as indicated by a bone mineral density of the lumbar vertebra and proximal femur of t<-2.0 as obtained from dual energy x-ray absorptiometry (DEXA), or a DEXA scan completed within the last year.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael L. Madigan, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Tech, Blacksburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Received no training.
Period: Overall Study
Arm/Group | Step Training | Treadmill Training | Control
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Step Training | Treadmill Training | Control | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (4.1) | 71.8 (5.2) | 71.8 (4.3) | 71.8 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 6 | 18
  Male | 4 | 4 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 9 | 10 | 29
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 9 | 10 | 10 | 29
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30
body height [Mean (Standard Deviation); unit: meters] | 1.63 (0.08) | 1.69 (0.10) | 1.70 (0.12) | 1.68 (0.10)
body mass [Mean (Standard Deviation); unit: kilograms] | 69.9 (17.0) | 79.6 (15.8) | 81.9 (16.8) | 77.1 (16.8)
unipedal stance time (seconds) [Mean (Standard Deviation); unit: seconds] | 18.9 (11.5) | 16.5 (12.7) | 17.3 (13.8) | 17.6 (12.3)

OUTCOME MEASURES:

1. Primary Outcome: Trunk Angle at Touchdown of the First Recovery Step
Description: After a laboratory-induced trip: Angle from vertical of a line connecting midpoint of greater trochanter markers and midpoint of the acromion markers
Time Frame: 1 week after the 3-week intervention
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: trips
Arm/Group | Step Training | Treadmill Training | Control
Number analyzed (Participants) | 10 | 10 | 10
Number analyzed (trips) | 10 | 10 | 10
degrees | 27.0 (8.2) | 24.6 (7.4) | 28.4 (6.9)

2. Primary Outcome: Trip Outcome
Description: This is a binary variable that has a value of either "fall" or "recovery."
  After a laboratory-induced trip, trip outcome will be assign to one of the following two values:
  "fall" if a participant is fully and continuously supported by the harness as observed from video, or if the harness force applied to the participant, integrated over time from trip onset until 1 second after touchdown of the first recovery step, is greater than 40% of body weight * seconds. The harness force will be measured by a uniaxial load cell.
  "recovery" if the harness force applied to the participant, integrated over time from trip onset until 1 second after touchdown of the first recovery step, is less than 40% of body weight * seconds. The harness force will be measured by a uniaxial load cell.
Time Frame: 1 week after the 3-week intervention
Measure: Number; unit: number of falls
Units Other Than Participants: trips
Arm/Group | Step Training | Treadmill Training | Control
Number analyzed (Participants) | 10 | 10 | 10
Number analyzed (trips) | 10 | 10 | 10
number of falls | 4 | 10 | 8

3. Secondary Outcome: Recovery Step Length
Description: After a laboratory-induced trip, the distance between a lateral malleolus marker of the stance limb and a lateral malleolus marker of the stepping foot at touchdown
Time Frame: 1 week after the 3-week intervention
Measure: Mean (Standard Deviation); unit: % body height
Units Other Than Participants: trips
Arm/Group | Step Training | Treadmill Training | Control
Number analyzed (Participants) | 10 | 10 | 10
Number analyzed (trips) | 10 | 10 | 10
% body height | 49.5 (9.9) | 45.4 (5.2) | 40.1 (6.2)

4. Secondary Outcome: Sacrum Height at Touchdown of the First Recovery Step
Description: After a laboratory-induced trip, the minimum distance between the walkway and the greater trochanter marker on the non-tripping limb during trip recovery.
Time Frame: 1 week after the 3-week intervention
Measure: Mean (Standard Deviation); unit: % of sacrum height while standing
Units Other Than Participants: trips
Arm/Group | Step Training | Treadmill Training | Control
Number analyzed (Participants) | 10 | 10 | 10
Number analyzed (trips) | 10 | 10 | 10
% of sacrum height while standing | 97.4 (7.3) | 96.7 (10.1) | 97.7 (13.0)

5. Secondary Outcome: Gait Speed
Description: The average forward speed of the participant prior to the laboratory-induced trip.
Time Frame: 1 week after the 3-week intervention
Measure: Mean (Standard Deviation); unit: meters per second
Units Other Than Participants: trips
Arm/Group | Step Training | Treadmill Training | Control
Number analyzed (Participants) | 10 | 10 | 10
Number analyzed (trips) | 10 | 10 | 10
meters per second | 1.6 (0.2) | 1.5 (0.2) | 1.5 (0.2)

6. Secondary Outcome: Average Step Speed
Description: After a laboratory-induced trip, the distance between a lateral malleolus marker of the stance limb and a lateral malleolus marker of the stepping foot at touchdown divided by the time from impact with the trip obstacle and touchdown of the initial recovery step.
Time Frame: 1 week after the 3-week intervention
Measure: Mean (Standard Deviation); unit: meters per second
Units Other Than Participants: trips
Arm/Group | Step Training | Treadmill Training | Control
Number analyzed (Participants) | 10 | 10 | 10
Number analyzed (trips) | 10 | 10 | 10
meters per second | 1.7 (0.4) | 1.6 (0.2) | 1.4 (0.3)

7. Secondary Outcome: Trip Recovery Strategy
Description: This is a binary variable that has a value of either "elevating" or "lowering."
  Elevating or lowering, depending upon how the participant uses the foot that trips on the obstacle after the laboratory-induced trip. If the foot is elevated over the obstacle, then this will be elevating. If the foot is lowered to the ground and the opposite foot first steps over the obstacle, then this will be lowering. The measurement tool to determine this outcome is a video recording of the trip, and this outcome has no units.
Time Frame: 1 week after the 3-week intervention
Measure: Number; unit: number of trips using lowering strategy
Units Other Than Participants: trips
Arm/Group | Step Training | Treadmill Training | Control
Number analyzed (Participants) | 10 | 10 | 10
Number analyzed (trips) | 10 | 10 | 10
number of trips using lowering strategy | 12 | 12 | 13

ADVERSE EVENTS:
Time Frame: 1 week after the 3-week intervention
Description: Definitions did not differ from clinicaltrials.gov
Arm/Group | Step Training | Treadmill Training | Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-24): https://cdn.clinicaltrials.gov/large-docs/43/NCT05734443/Prot_SAP_000.pdf
  • Informed Consent Form (2025-03-24): https://cdn.clinicaltrials.gov/large-docs/43/NCT05734443/ICF_001.pdf